CLINICAL TRIAL: NCT01873560
Title: Influence of Fractional Flow Reserve (FFR) on the Clinical OutcomEs of PERcutaneouS Coronary Intervention (PCI): A ProspECTIVE, Multicenter FFR Registry
Brief Title: Influence of FFR on the Clinical Outcome After Percutaneous Coronary Intervention
Acronym: PERSPECTIVE
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Collaborators: Seoul National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Ulsan University Hospital (Other); Busan Veterans General Hospital (Unknown); Samsung Medical Center (Other); Sejong General Hospital (Other); Tokyo Medical University (Other); Gifu Heart Center (Other); Japanese Red Cross Kyoto Daini Hospital (Unknown)
Responsible Party: Principal Investigator, Joon Hyung Doh, Associate professor, Inje University
Other Study IDs: IB-2-1306-020
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Coronary Disease
Keywords: fractional flow reserve; drug eluting stent; coronary atherosclerosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FFRpost: High FFRpost group and low FFRpost group were defined according to the optimal cut-off value for predicting clinical outcome.

SUMMARY:
Fractional flow reserve (FFR) is a physiologic index for the determination of ischemia-causing coronary stenosis as well as drug eluting stent (DES) optimization, even multiple anatomic imaging parameters have been widely used in clinical practice for the assessment of optimal stent procedure. Prognostic value of post-stent FFR (FFRpost) have been rarely evaluated in patient treated with 2nd generation DES. This multicentre, prospective registry was aimed to evaluate the influence of physiologic parameters on the clinical outcome after 2nd generation DES implantation.

DETAILED DESCRIPTION:
Patients who diagnosed obstructive coronary artery disease and treated by DES with FFR examination would be enrolled, consecutively. FFR measurement would be required at the baseline and at the end of index PCI procedure. PCI procedure would be performed upon local routine. Any available 2nd generation DES could be used. Informed consent should be obtained and protocol should be approved by each collaborator's institutional review board (IRB). Web-based electronic-case record form (CRF) system will be used for collecting data. All data will be handled and analyzed by blind fashion at independent core lab. Patient will be followed-up at each collaborator's hospital at least 2 year after index procedure. Any adverse event will be reported and addressed immediately by appropriate medical treatment to protect patient.

ELIGIBILITY:
Inclusion Criteria:

* any patient meets eligible criteria who underwent PCI with DES followed by FFR measurement at the index procedure
* patient who provide informed consent

Exclusion Criteria:

* culprit vessel of acute coronary syndrome
* failed achieving TIMI 3 flow at the end of PCI
* left ventricular ejection fraction <30%
* graft vessel
* collateral feeder
* in-stent stenosis
* primary myocardial or valvular heart disease
* in patient whose life expectancy less than 2 years
* visible thrombus of target vessel segment

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed obstructive coronary artery disease and treated by DES with FFR examination at the index procedure
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2013-05; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Target-vessel failure | 2 years after index procedure
  During two-year follow-up period, target-vessel failure (composite of cardiac death, target-vessel related myocardial infarction, and clinically-driven target vessel revascularization) will be evaluated. Target vessel will be defined as the treated vessel with DES which assessed by post-stent FFR.
  All clinical outcome will be reported according to the location of target vessel (LAD vs. non-LAD).

SECONDARY OUTCOMES:
clinical, angiographic and physiologic predictors for target-vessel failure | 2 years after index procedure
  Clinical, angiographic and physiologic predictors for target-vessel failure by univariate and multivariate analysis will be performed.

OTHER OUTCOMES:
Intravascular ultrasound (IVUS) derived predictors for post-stent FFR and target vessel failure | 2 years after index procedure
  In patient who performed IVUS examination, IVUS derived parameters will be evaluated for the prediction of post-stent FFR and target-vessel failure

CONTACTS AND LOCATIONS:
Overall Officials: Joon Hyung Doh, MD, PhD, Principal Investigator — Inje Univesity Ilsan Paik Hospital; Bon-Kwon Koo, Study Director — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Background] Pijls NH, Klauss V, Siebert U, Powers E, Takazawa K, Fearon WF, Escaned J, Tsurumi Y, Akasaka T, Samady H, De Bruyne B; Fractional Flow Reserve (FFR) Post-Stent Registry Investigators. Coronary pressure measurement after stenting predicts adverse events at follow-up: a multicenter registry. Circulation. 2002 Jun 25;105(25):2950-4. doi: 10.1161/01.cir.0000020547.92091.76. PMID 12081986
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Nam CW, Hur SH, Cho YK, Park HS, Yoon HJ, Kim H, Chung IS, Kim YN, Kim KB, Doh JH, Koo BK, Tahk SJ, Fearon WF. Relation of fractional flow reserve after drug-eluting stent implantation to one-year outcomes. Am J Cardiol. 2011 Jun 15;107(12):1763-7. doi: 10.1016/j.amjcard.2011.02.329. Epub 2011 Apr 8. PMID 21481828
- [Background] Samady H, McDaniel M, Veledar E, De Bruyne B, Pijls NH, Fearon WF, Vaccarino V. Baseline fractional flow reserve and stent diameter predict optimal post-stent fractional flow reserve and major adverse cardiac events after bare-metal stent deployment. JACC Cardiovasc Interv. 2009 Apr;2(4):357-63. doi: 10.1016/j.jcin.2009.01.008. PMID 19463450
- [Derived] Lee HJ, Mejia-Renteria H, Escaned J, Doh JH, Lee JM, Hwang D, Yuasa S, Choi KH, Jang HJ, Jeon KH, Lee J, Nam CW, Shin ES, Koo BK. Prediction of functional results of percutaneous coronary interventions with virtual stenting and quantitative flow ratio. Catheter Cardiovasc Interv. 2022 Dec;100(7):1208-1217. doi: 10.1002/ccd.30451. Epub 2022 Nov 2. PMID 36321601
- [Derived] Lee SH, Kim J, Lefieux A, Molony D, Shin D, Hwang D, Choi KH, Chang HS, Jeon KH, Lee HJ, Jang HJ, Kim HK, Ha SJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Doh JH, Shin ES, Nam CW, Koo BK, Gwon HC, Lee JM. Clinical and Prognostic Impact From Objective Analysis of Post-Angioplasty Fractional Flow Reserve Pullback. JACC Cardiovasc Interv. 2021 Sep 13;14(17):1888-1900. doi: 10.1016/j.jcin.2021.07.014. PMID 34503739
- [Derived] Shin D, Dai N, Lee SH, Choi KH, Lefieux A, Molony D, Hwang D, Kim HK, Jeon KH, Lee HJ, Jang HJ, Ha SJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Doh JH, Shin ES, Nam CW, Koo BK, Gwon HC, Ge J, Lee JM. Physiological Distribution and Local Severity of Coronary Artery Disease and Outcomes After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2021 Aug 23;14(16):1771-1785. doi: 10.1016/j.jcin.2021.06.013. PMID 34412795
- [Derived] Hwang D, Lee JM, Lee HJ, Kim SH, Nam CW, Hahn JY, Shin ES, Matsuo A, Tanaka N, Matsuo H, Lee SY, Doh JH, Koo BK. Influence of target vessel on prognostic relevance of fractional flow reserve after coronary stenting. EuroIntervention. 2019 Aug 29;15(5):457-464. doi: 10.4244/EIJ-D-18-00913. PMID 30561367
- [Derived] Lee JM, Hwang D, Choi KH, Rhee TM, Park J, Kim HY, Jung HW, Hwang JW, Lee HJ, Jang HJ, Kim SH, Song YB, Cho YK, Nam CW, Hahn JY, Shin ES, Kawase Y, Matsuo A, Tanaka N, Doh JH, Koo BK, Matsuo H. Prognostic Implications of Relative Increase and Final Fractional Flow Reserve in Patients With Stent Implantation. JACC Cardiovasc Interv. 2018 Oct 22;11(20):2099-2109. doi: 10.1016/j.jcin.2018.07.031. PMID 30336814